CLINICAL TRIAL: NCT06271551
Title: Transdermal Estradiol and Exercise in Mitigating Adverse Effects of Androgen Deprivation Therapy for Prostate Cancer Radiation Therapy: A Randomized Controlled Trial
Brief Title: Transdermal Estradiol and Exercise in Mitigating Adverse Effects of Androgen Deprivation Therapy for Prostate Cancer Radiation Therapy
Acronym: ESTRACISE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Collaborators: Tampere University (Other); University of Jyvaskyla (Other); Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESTRACISE
Record Dates: First submitted 2023-11-20; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 fashion to receive transdermal estradiol and androgen deprivation or solely androgen deprivation therapy. In addition subgroup of participants are randomized in a 1:1 fashion to perform resistance training or to be allocated in non-training control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdermal estradiol (Experimental): Participants (n=155) receiving transdermal estradiol and androgen deprivation therapy.
  Interventions: Drug: Transdermal estrogen; Behavioral: Resistance training
- Androgen deprivation therapy (Active Comparator): Participants (n=155) receiving solely androgen deprivation therapy.
  Interventions: Drug: Active Comparator: Androgen deprivation therapy; Behavioral: Resistance training

INTERVENTIONS:
Drug: Transdermal estrogen — Participants (n=155) receiving transdermal estradiol for 12 months.
  Arms: Transdermal estradiol
Drug: Active Comparator: Androgen deprivation therapy — Participants (n=155) receiving solely androgen deprivation therapy for 12 months.
  Arms: Androgen deprivation therapy
Behavioral: Resistance training — Participants (n=30 in each arm) performing supervised resistance training for six months.

SUMMARY:
The goal of the clinical trial is to find out whether transdermal estradiol will reduce the adverse effects of androgen deprivation therapy in prostate cancer patients.

The primary aim of this study is to estimate the efficacy of transdermal estradiol (E2) in reducing androgen deprivation therapy induced adverse effects on sexual function. A secondary aim of this study is to estimate the utility of E2 and the combination of E2 with supervised exercise in reducing other androgen deprivation therapy related adverse effects.

Participants (n=310) will use transdermal estradiol for 12 months concomitant to androgen deprivation therapy. The use of transdermal estradiol will start at the beginning of the trial, at the same time as androgen deprivation therapy. A subgroup of participants (n=120) will also be allocated to perform six months supervised resistance training.

Researchers will compare transdermal estradiol group to control group, and resistance training groups and non-training control groups.

DETAILED DESCRIPTION:
The current study is an open-label study examining a drug with known tolerability and safety profile (phase IIA trial). The study will recruit 310 prostate cancer patients with high-risk disease and scheduled for external beam radiation with adjuvant subcutaneous androgen deprivation therapy, leuprorelin (LHRH agonist).

Stratified randomization (n=310) will be done in a 1:1 fashion to the transdermal estradiol + androgen deprivation therapy arm or control arm (androgen deprivation therapy only). Stratified randomization will be based on two covariates, which are sexual dysfunction score and BMI. The use of the stratified randomization method will guarantee even distribution of covariates, which could likely affect the study outcomes. Additionally, a total of 120 participants who are willing to participate in the supervised resistance training program and have sufficient performance status (ECOG 0-1) will be randomized to the resistance training group or the non-training control group. A total of 30 men from each arm will be recruited to supervised training and 30 men from each arm the non-training control group. Participants of the ESTRACISE who do not participate in the exercise substudy will form a non-training group (n=95 per arm). The stratified randomization of the substudy participants in the training group or the non-training control group will be done in a 1:1 fashion before the start of the training period. Stratified randomization will be based on two main covariates, which are age and the self-reported physical activity level of the participant.

ESTRACISE participants allocated to the transdermal estradiol arm will use transdermal estradiol gel (E2) as a dose of 750 ug (EstroGel 0.6 mg/ml) in addition to androgen deprivation therapy for 12 months. Additionally, substudy participants allocated to the resistance training groups will be attending supervised group resistance training sessions twice a week for six months. The resistance training will start after six months of androgen deprivation therapy. Participants in the non-training groups are advised to stay physically active but they will do it at their own discretion.

According to the standard treatment protocol, all participants will receive androgen deprivation therapy as leuprorelin, subcutaneous injections at three months intervals for a minimum of one year, and standard external beam radiation for prostate cancer with standard clinical dosing and fractionation at the discretion of the radiation oncologist.

The research methodologies include questionnaires (expanded prostate cancer index composition 26, world health organization quality of life brief version, and patient health questionnaire), adverse event screening, medication compliance screening, computerized tomography (CT) of the thigh muscle, bioimpedance analysis (BIA), 3D-imaging of the body composition, body composition and bone mineral assessment by dual-energy x-ray absorptiometry (DXA), strength, functional capacity, physical activity measurements, and serum and plasma blood samples. In addition, muscle biopsies are collected from a subset of participants allocated in the resistance training (n=60) and non-training control groups (n=60). The primary measurement timepoints are baseline (0 months), after six months of androgen deprivation therapy, and after twelve months of androgen deprivation therapy.

Based on prior sample size estimation of primary outcome the n=310 should be more than adequate to detect statistically significant differences in the mean sexual domain score between the two study arms. The true difference in the mean is expected to be 10, with a probability (power) of 0.8, a Type 1 error probability of 0.05, and with dropout rate of 10%.

ELIGIBILITY:
Inclusion Criteria:

* Men with localized prostate cancer, and scheduled for external beam radiation with adjuvant subcutaneous androgen deprivation therapy, leuprorelin (LHRH agonist) for at least 12 months without any other endocrinology treatments for prostate cancer
* Adults (age over 18 years)
* Sufficient performance status (Eastern Cooperative Oncology Group, 0-1)
* Body mass index between 18.5 - 30.0
* Willingness to participate and signed consent

Exclusion Criteria:

* Patients with low-risk prostate cancer (ISUP Gleason grade 1)
* Patients with expected adjuvant androgen deprivation therapy for less than one year
* Distant bone, lymph node, or soft tissue metastasis
* Cardiac pacemaker
* Prior recent cardiovascular event or stroke (<12 months)
* Past or current venous thromboembolism
* Other untreated or unstable malignancy in risk of recurrence/progression (as judged by the treating physician)
* Concurrent glucocorticoid treatment
* Physical disabilities for regular exercise
* Any medication or condition considered as a contraindication to estradiol (allergy to adjuvant compounds (carbomer, trolamine), history with thromboembolic disorders (protein C, protein S, or antithrombin deficiency), porphyria, acute or previous liver disease, drugs with cytochrome P450 enzyme metabolism (anticonvulsants: phenobarbital, phenytoin, carbamazepine; anti-infectives: rifampicin, rifapentine, nevirapine, efavirenz; and St. John's wort)) or leuprorelin (allergy to adjuvant compounds (polylactic acid), Qt-time prolonging drugs (quinidine, disopyramide, amiodarone, sotalol, dofetilide, ibutilide, methadone, moxifloxacin, antipsychotics)
* Known allergy to estradiol or leuprorelin
* Expected poor compliance or expected survival time of less than one year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of transdermal estradiol in mitigating the deterioration of EPIC-26 (The Expanded Prostate Cancer Index Composite) sexual function domain scores caused by androgen deprivation therapy. | Twelve and six months.
  Compared between the two arms. Scores scaled from 0 - 100, higher score means better sexual function.

SECONDARY OUTCOMES:
The occurrence of androgen deprivation therapy induced adverse effects. | Twelve and six months.
  Compared between different groups. Assessed by CTCAE (Common Termionology Criteria for Adverse Events). Number of participants with androgen deprivation therapy related adverse events, and grading of adverse event from 1 - 5. Higher grading indicates worse adverse event.
Number of participants with transdermal estradiol-related adverse events as assessed by CTCAE (Common Terminology Criteria for Adverse Events). | Twelve and six months.
  Transdermal estradiol arm. Number and grading of adverse events from 1 - 5. Higher grading means worse adverse event.
Impact of transdermal estradiol with or without 6-month supervised resistance training on one repetition maximum tests of both the leg press and barbell biceps curl, and maximal hand grip strength assessed with a dynamometer. | Twelve and six months.
  Compared between different groups. One repetition maximum tests and maximal hand grip strength assessed as kilograms or newtons. Higher kilograms or newtons indicates higher strength.
Impact of transdermal estradiol with or without 6-month supervised resistance training on explosive strength of the leg extensors assessed with a countermovement jump (CMJ). | Twelve and six months.
  Compared between different groups. From CMJ flight time is defined as milliseconds. Higher flight time in milliseconds represents higher jump height and explosive strength.
Impact of transdermal estradiol with or without 6-month supervised resistance training on 6-minute walk (functional capacity). | Twelve and six months.
  Compared between different groups. Walking distance and heart rate will be collected from 6-minute walk test. Higher walking distance with lower heart rate indicates better functional capacity.
Impact of transdermal estradiol with or without 6-month supervised resistance training on loaded 10-stair climb test (functional capacity). | Twelve and six months.
  Compared between different groups. Time taken to ascend and descend from 10-stair climb test. Less time taken to complete 10-stair climb test indicates better functional capacity.
Impact of transdermal estradiol with or without 6-month supervised resistance training on body composition. | Twelve and six months.
  Compared between different groups. More lean mass, and less fat mass indicates better body composition.
Impact of transdermal estradiol with or without 6-month supervised resistance training on bone mineral density. | Twelve and six months.
  Compared between different groups. Higher bone mineral density indicates better outcome.
Impact of transdermal estradiol with or without 6-month supervised resistance training on mid-thigh muscle mass. | Twelve and six months.
  Compared between different groups. Higher mid-thigh muscles cross-sectional area indicates higher mid-thigh muscle mass.
Impact of transdermal estradiol with or without 6-month supervised resistance training on mid-thigh fat mass. | Twelve and six months.
  Compared between different groups. Lower adipose tissue size indicates less mid-thigh fat mass.
Impact of transdermal estradiol with or without 6-month supervised resistance training on hormone (testosterone and estradiol) levels, and cancer (PSA) status. | Twelve and six months.
  Compared between different groups. Higher or lower hormones levels could indicate better outcome, depending on the arm of the participant, and overall status. Lower PSA concentration usually indicates better outcome.
Impact of transdermal estradiol with or without 6-month supervised resistance training on concentration of PVK, IL-6, TNF-α, AFOS, Alat, Krea, Cholesterol, LDL-C, HDL-C, and triglycerides). | Twelve and six months.
  Compared between different groups. Higher or lower concentration of biomarkers can indicate better outcome, depending on the exact biomarker.
Impact of transdermal estradiol with or without 6-month supervised resistance training on type I and II myofibers' cross-sectional area, myonuclei, myonuclear domain, the satellite cell count, androgen receptor and myostatin content | Twelve and six months.
  Compared between different groups. Higher type I and II myofibers' cross-sectional area indicates improved skeletal muscle characteristics. Higher myonuclei, myonuclear domain, satellitte cell count, and androgen and myostatin content usually indicates improved cellular function.
Impact of transdermal estradiol with or without 6-month supervised resistance training on muscle cellular function (e.g., HSP70, alpha B-crystallin, HSP60, cytochrome c oxidase subunit IV proteins) | Twelve and six months.
  Compared between different groups. Higher or lower concentration of proteins could indicate improved or worsen muscle cellular function, depending on the exact protein.
Number of participants with resistance training induced adverse events. | Twelve and six months.
  Compared between different groups. Assessed by CTCAE (Common Termionology Criteria for Adverse Events). Number of participants with androgen deprivation therapy related adverse events, and grading of adverse event from 1 - 5. Higher grading indicates worse adverse event.
The World Health Organization Quality of Life Brief Version (WHOQOL-BREF). | Twelve and six months.
  Compared between different groups. Subdomain scores scaled from 0 to 100. Higher overall and subdomain score in WHOQOL-BREF indicates higher quality of life.
The Patient Health Questionnaire score (PHQ-9) overall and subdomain score. | Twelve and six months.
  Compared between different groups. Scores scaled from 0 to 27. Higher overall score in PHQ-9 indicates more depressive symptoms.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jussila I, Ahtiainen JP, Laakkonen EK, Siltari A, Kaipia A, Jokela T, Karkkainen M, Newton R, Raastad T, Huhtala H, Murtola TJ, Seikkula H. Transdermal oestradiol and exercise in androgen deprivation therapy (ESTRACISE): protocol. BJU Int. 2024 Jul;134(1):110-118. doi: 10.1111/bju.16361. Epub 2024 Apr 8. PMID 38587276